CLINICAL TRIAL: NCT02780349
Title: Evaluation of WIRION™ EPS in Lower Extremities Arteries
Acronym: WISE-LE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Gardia Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CL-003
Record Dates: First submitted 2016-05-19; First posted 2016-05-23 (Estimated); Results first posted 2018-02-14 (Actual); Last update posted 2018-03-15 (Actual); Status verified 2018-02

CONDITIONS: Peripheral Arterial Disease (PAD)
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- WIRION EPS (Experimental): Single arm study. All patients undergo procedure with the WIRION EPS
  Interventions: Device: WIRION

INTERVENTIONS:
Device: WIRION — Embolic Protection System

SUMMARY:
Demonstrate the safety and performance of the WIRION™ EPS in subjects undergoing lower extremity atherectomy for the treatment of Peripheral Arterial Disease (PAD)

ELIGIBILITY:
Inclusion Criteria:

1. Subject is at least 18 years of age
2. Subject or authorized representative, signed a written Informed Consent form to participate in the study, prior to any study related procedures
3. Subject is willing to comply with the protocol requirements and return to the treatment center for all required clinical evaluations
4. Rutherford classification 2-4
5. Has moderate to severe calcification visualized on angiogram in the femoropopliteal arteries
6. Planned atherectomy of the native femoropopliteal arteries
7. Reference vessel diameter for intended filter location must be visually estimated to be ≥3.5mm and ≤6.0mm
8. An adequate "landing zone" for placement of the WIRION™ device distal to the target lesion of at least 30mm
9. A female subject is eligible if not of child bearing potential or has a negative pregnancy test within the previous 7 days and agrees to remain on birth control throughout the study

Exclusion Criteria:

1. Any planned surgical or endovascular intervention within 30 days before or after the index procedure
2. A lesion deemed not accessible by the WIRION™ EPS
3. Inability to take aspirin or ADP receptor antagonists
4. History of bleeding diathesis or coagulopathy or will refuse blood transfusion if deemed necessary
5. Has perforation, dissection, or other injury of the access or target vessel requiring additional stenting or surgical intervention before enrollment
6. Subject is enrolled in another drug or device study protocol that has not reached its primary endpoint (participating in registry studies is not excluded)
7. Life expectancy less than 12 months
8. Known severe renal insufficiency (eGFR <30 ml/min/1.72m2).
9. ≤1-vessel tibial run-off status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 103 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William Gray, MD, Principal Investigator — Main Line Health
Locations (10):
- United States (8):
  - Denver VA Medical Center, Denver, Colorado
  - Unity Point, Davenport, Iowa
  - Ochsner Clinic, New Orleans, Louisiana
  - St Elizabeth Medical Center, Boston, Massachusetts
  - St John Hospital, Detroit, Michigan
  - Columbia Presbyterian, New York, New York
  - Lankenau Institute for Medical Research, Philadelphia, Pennsylvania
  - Miriam Hospital, Providence, Rhode Island
- Germany (2):
  - Universitats herzzentrum Bad Krozingen, Bad Krozingen
  - Universitatklinikum Leipzig, Leipzig

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | WIRION EPS
Started | 103
Completed | 101
Not Completed | 2

BASELINE CHARACTERISTICS:
Groups:
- Single Arm: WIRION: Embolic Protection System
Arm/Group | Single Arm
Number analyzed (Participants) | 103
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.2 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32
  Male | 71
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 93
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 79
  Germany | 24

OUTCOME MEASURES:

1. Primary Outcome: Freedom From Major Adverse Events (MAE) to 30 Days Post Procedure.
Description: MAE defined as a serious adverse event that results in death, acute myocardial infarction, thrombosis, pseudo-aneurysm, dissection (grade C or greater) or clinical perforation at the filter location, distal embolism (clinically relevant), unplanned amputation, or clinically-driven target vessel revascularization (TVR), through 30 days post-procedure, as adjudicated by the Clinical Events Committee (CEC)
Time Frame: 30 days
Measure: Count of Participants; unit: Participants
Arm/Group | Single Arm
Number analyzed (Participants) | 103
Participants | 2

ADVERSE EVENTS:
Time Frame: 30 days follow up period
Arm/Group | Single Arm
All-Cause Mortality (participants affected / at risk) | 0/103
Serious Adverse Events (participants affected / at risk) | 8/103
Other Adverse Events (participants affected / at risk) | 9/103
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=103)
Hypotension, Hemoglobin drop (Cardiac disorders) | 1
Access site complication (Vascular disorders) | 1
Vessel occlusion (Vascular disorders) | 1
TVR (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 3
Dyspenea (Cardiac disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Single Arm (N=103)
Dissection (Vascular disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-20): https://cdn.clinicaltrials.gov/large-docs/49/NCT02780349/Prot_SAP_000.pdf